CLINICAL TRIAL: NCT04738526
Title: One Year Clinical Evaluation of Shade Matching and Patient Satisfaction of New Gradient Technology Monolithic Zirconia (5Y-TZP\3Y-TZP) Compared to Lithium Disilicate Crowns in Dental Esthetic Zone (Randomized Clinical Trial)
Brief Title: One Year Clinical Evaluation of Shade Matching and Patient Satisfaction of New Gradient Technology Monolithic Zirconia (5Y-TZP\3Y-TZP) Compared to Lithium Disilicate Crowns in Dental Esthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Khaled Abd El Kader Eid, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 361020
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Decayed Teeth; Malposed Teeth; Endodontically Treated Teeth; Teeth Restored With Large Filling Restorations; Single Anterior Crowns; Single Premolars Crowns
MeSH Terms: conditions — Dental Caries; Tooth, Nonvital | interventions — lithia disilicate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- natural tooth (Active Comparator)
  Interventions: Other: natural tooth
- lithium disilicate (IPS e-max) ceramic crown (Experimental): monolithic lithium disilicate (IPS e-max) ceramic crown for crowns in esthetic zone
  Interventions: Other: lithium disilicate (IPS e-max) ceramic crown
- New gradient technology zirconia (5Y-TZP\ 3Y-TZP) IPS e.max ZirCad Prime ceramic crown (Experimental)
  Interventions: Other: New gradient technology zirconia (5Y-TZP\ 3Y-TZP) IPS e.max ZirCad Prime ceramic crown

INTERVENTIONS:
Other: lithium disilicate (IPS e-max) ceramic crown — monolithic lithium disilicate ceramic crown
  Arms: lithium disilicate (IPS e-max) ceramic crown
Other: New gradient technology zirconia (5Y-TZP\ 3Y-TZP) IPS e.max ZirCad Prime ceramic crown — conjunction with the two zirconium oxide raw materials 3Y-TZP and 5Y-TZP is responsible for producing a continuous, seamless progression of the shade and translucency within the material
  Arms: New gradient technology zirconia (5Y-TZP\ 3Y-TZP) IPS e.max ZirCad Prime ceramic crown
Other: natural tooth — natural tooth is composed of enamel. Enamel is on the surface of every tooth and it has a natural hue of white. However, the underlying dentin layer has a slightly yellowish color. This yellowish hue shows through the enamel in almost everyone
  Arms: natural tooth

SUMMARY:
Although zirconia is widely used for fabrication of restorations, the 3Y-TZP zirconia where limited for posterior region for its high strength and bad esthetic. While the 5Y-TZP zirconia is limited for the anterior region due to its good esthetic and low strength. For that reason, the introduction of the new gradient technology zirconia (5Y-TZP\3Y-TZP) (IPS e.max Zircad Prime) has offered a solution to solve this problem be combining the esthetic of 5Y-TZP and the high strength of 3Y-TZP. The aim of the present study is to evaluate shade matching to natural tooth and patient satisfaction of the new gradient technology zirconia (5Y-TZP\3Y-TZP) and lithium disilicate ceramic crowns.

DETAILED DESCRIPTION:
Restorative dentistry is a mix of science and art. The success of restorative dentistry is determined on the basis of functional and esthetic results. Closely matching natural teeth with an artificial restoration can be one of the most challenging procedures in restorative dentistry. Natural teeth vary greatly in color and shape.The color of a ceramic restoration is affected by the shade of the ceramic material, its thickness, and, the color of the underlying material. The restoration's color is influenced by ceramic firing temperature, the color of the prepared tooth, translucency and thickness of veneering porcelain.

The rational of this study is newly introduced gradient technology zirconia (5Y-TZP\3Y-TZP) (IPS e.max Zircad Prime) with improved optical properties to solve the drawbacks of esthetic properties of zirconia.

Null hypothesis of the study will be:

* There would be no difference in shade matching of the new gradient technology zirconia (5Y-TZP\3Y-TZP) and lithium disilicate ceramic crowns used in the esthetic zone.
* There would be no difference in patient satisfaction of new gradient technology zirconia (5Y-TZP\3Y-TZP) and lithium disilicate ceramic crowns at baseline, 3, 6, 9, 12 months used in the esthetic zone.

ELIGIBILITY:
Inclusion Criteria:

1. From 21-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations.
3. Psychologically and physically able to withstand conventional dental procedures.
4. Patient with thick gingival biotype.
5. Patients with teeth problems indicated for single all ceramic restoration in esthetic zone

   1. Badly decayed teeth.
   2. Teeth restored with large filling restorations.
   3. Endodontically treated teeth.
   4. Malformed teeth.
   5. Malposed teeth (Tilted, over-erupted, rotated, etc.).
   6. Spacing between teeth in esthetic zone.
6. Able to return for follow-up examinations and evaluation.

Exclusion Criteria:

1. Patient less than 21 or more than 50 years.
2. Patient with active resistant periodontal diseases.
3. Patients with poor oral hygiene and uncooperative patients.
4. Pregnant women.
5. Patients in the growth stage with partially erupted teeth.
6. Psychiatric problems or unrealistic expectations.
7. Patient with periodontal problems.
8. Patients with malocclusion or parafunctional habits.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
shade match | 1 year
  measured by Modified United States Public Health Service criteria (USPHS criteria) Score Alpha(A):matches tooth Bravo(B):acceptable mismatch Charlie(C):unacceptable mismatch

SECONDARY OUTCOMES:
Shade match | 1 year
  measured by Vita Easyshade V spectrophotometer

OTHER OUTCOMES:
Patient satisfaction | 1 year
  measured by Visual Analog Scale Questionnaire (VAS Questionnaire) ("0" unsatisfied - "10" satisfied)

IPD SHARING:
Plan to Share IPD: Undecided